CLINICAL TRIAL: NCT01987271
Title: Effects Of Noninvasive Ventilation During The Treadmill Walking Test On Cardiorespiratory System, Walk Distance, And Thoracoabdominal Kinematics Of Patients With Cystic Fibrosis: Clinical Randomized Controlled Trial.
Brief Title: Effects Of Noninvasive Ventilation On Functional Capacity Of Patients With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Cibelle Andrade Lima, Master - Universidade Federal de Pernambuco, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0.381.0.172.099-11
Record Dates: First submitted 2013-11-04; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Cystic Fibrosis
Keywords: exercise tolerance; exercise test; noninvasive ventilation
MeSH Terms: conditions — Cystic Fibrosis | interventions — Noninvasive Ventilation; Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With noninvasive ventilation (Experimental): When patients do the six minute walk test with the noninvasive ventilation.
  Interventions: Device: Noninvasive Ventilation
- Without noninvasive ventilation (No Intervention): When patients do the six minute walk test without noninvasive ventilation.

INTERVENTIONS:
Device: Noninvasive Ventilation — A randomized plan define the order in which patients would execute the 6MWT, with or without NIV.
  Other Names: BiLEVEL; Noninvasive ventilatory support
  Arms: With noninvasive ventilation

SUMMARY:
The purpose of this study is to evaluate the effect of noninvasive ventilation (NIV) in functional capacity of children and adolescents with cystic fibrosis.

DETAILED DESCRIPTION:
This is an open randomized controlled crossover clinical trial. Sample selection was by convenience and patients were screened at the Pneumology outpatient facility of the Instituto de Medicina Integral Professor Fernando Figueira (IMIP) in Recife, Brazil.

The sample was calculated using a software developed by the MGH Mallinckrodt General Clinical Research Center, based on the results of the first 10 volunteers, for a statistical power of detecting differences between procedures of 80% and a significance level of 0.05. A sample size of n=13 patients was determined, considering that the real difference between the walk distance between procedures with and without NIV is 0.03 km and the standard deviation of the differences in variables is 0.034 km.

All patients agreed to take part in the study by giving their informed consent, in accordance with resolution 196/96 of the National Health Council.

Technical Procedures Patients were initially assessed for current and past conditions, medication use and anthropometric data (height, weight and body mass index - BMI). Next, a randomized plan was compiled using the Web Site Randomization.com, applying a generator of random-permuted blocks to define the order in which patients would execute the 6MWT, with or without NIV. Patients allocated to group 1 (G1) initiated the 6MWT without NIV to subsequently perform the test with ventilatory support, since those allocated to group 2 (G2) underwent the tests in reverse order. A minimum and maximum rest period of 24 and 48 hours, respectively, was observed between tests.

Before and after the 6MWT with and without NIV, patients were assessed for variations in compartmental chest wall volume and ventilatory pattern by optoelectronic plethysmography (OEP), which was followed by the spirometric test. A 20-minute rest period was given after the pulmonary function test before proceeding to the 6MWT.

6-minute walk test on the treadmill: Prior to the test, the patient was familiarized with the treadmill (G-635, Pro Action BH-fitness- Germany) and instructed about test procedures in accordance with ATS guidelines22. The following parameters were assessed before, immediately after and in the 5th minute post-test: blood pressure (BP), respiratory rate (RR), heart rate (HR), Borg's scale (BS) and peripheral O2 saturation (SpO2). HR, RR and SpO2 were also monitored minute by minute during the test, such that a drop in SpO2 below 87% or rise in RR to more than 75% of age-predicted maximal HR were used as criteria for interrupting the test. The test initiated with the treadmill traveling at 2.5 km/h. Every 30 seconds of the test, the examiner asked the patient if the speed could be increased, maintained or decreased, and patients answered using previously agreed upon signals. The speed could not exceed 7 km/h and if it was reached, the question would be re-asked in the next 30 seconds to determine whether the speed would be maintained or reduced. After the test, the walk distance (WD) on the treadmill was recorded.

The 6MWT performed with NIV followed the same procedures described above. However, before the test, patients were submitted to NIV on a BiPAP mode (Synchrony- Respironics, Brazil) for 30 minutes, as proposed by Serra et al 15, with inspiratory airway pressure (IPAP) level of 12 cmH2O and final expiratory airway pressure (EPAP) of 6 cmH2O, which can vary by 2 cmH2O more or less depending on the patient's comfort. In the last six minutes of BiPAP the patient performed the 6MWT with the ventilatory support.

Optoelectronic plethysmography: The individual was sitting with 89 retro-reflective sensors at specific thoracic and abdominal points. Eight cameras were arranged around the patient for a three-minute film of quiet breathing. The images were analyzed in a three-dimensional polyhedric model using OEP capture software (BTS Bioengineering, Italy). The following variables were assessed by OEP (BTS Bioengineering, Italy) before and after both tests, with and without NIV: tidal volume, pulmonary rib cage volume, abdominal rib cage and abdominal volume (VC, Vrcp Vrca, Vab), respiratory rate (RR), inspiratory time (Ti), expiratory time (Te) total ventilatory cycle time (Ttot) and duty cycle, which represents the Ti/Ttot ratio.

Spirometry: Spirometry was conducted using a Microloop MK 8 spirometer (Micro Medical, England) to assess pulmonary function response, considering a 20-minute rest period between the spirometric test and 6MWT. Three reproducible forced maneuvers that met American Thoracic Society criteria were performed. The highest values obtained for forced expiratory volume in the first minute (FEV1), forced vital capacity (FVC), forced vital capacity between 25-75% of FVC (FEF 25-75) were recorded for analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Cystic Fibrosis
* FEV1< 80% of predicted
* age between 7 and 16 years
* clinically stable patients
* no history of hospitalization for respiratory failure in the last three months

Exclusion Criteria:

* recent history of hemoptysis
* pneumothorax or evidence of emphysomatous bubbles detected by chest X-ray
* Burkholderia cepacia colonization
* the need for more than two physiotherapy sessions per day
* gastroesophageal reflux
* orthopedic trauma or cardiovascular conditions that impede the treadmill walk test
* heart failure

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Walk Distance (WD) on six minute walk test (6MWT) | 2 days
  Patients allocated to group 1 (G1) initiated the 6MWT without noninvasive ventilation (NIV) to subsequently perform the test with ventilatory support, since those allocated to group 2 (G2) underwent the tests in reverse order. Rest period between tests: 24 - 48 hours. At the end of the test, the walk distance on a treadmill is recorded.

SECONDARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | 2 days
  The patients do the walk test a twice on a week. Before and after each test, this variable is recorded.
Rib cage volumes | 2 days
  This variable is assessed by Optoeletronic Pletismography (BTS Bioengineering, Italy) before and after both tests, with and without NIV, recording the tidal volume, pulmonary rib cage volume, abdominal rib cage and abdominal volume (Vt, Vrcp Vrca, Vab).
Forced vital capacity (FVC) | 2 days
  The patients do the walk test a twice on the same week. Before and after each test, this variable is recorded.
Forced expiratory flow of 25% to 75% of FVC (FEF 25-75) | 2 days
  The patients do the walk test a twice on the same week. Before and after each test, this variable is recorded.
Respiratory cicle time | 2 days
  This following variable is assessed by Optoeletronic Pletismography (BTS Bioengineering, Italy) before and after both tests, with and without NIV, recording the respiratory rate (RR), inspiratory time (Ti), expiratory time (Te), total ventilatory cycle time (Ttot) and duty cycle, which represents the Ti/Ttot ratio.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Medicina Intergral Prof. Fernando Fiqueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Engelsbel S, Kuijper EJ, Dankert J, Braat MC, Egas J. [A tuberculosis project in Ecuador]. Ned Tijdschr Geneeskd. 1991 Dec 21;135(51):2428-32. Dutch. PMID 1758504
- [Result] Aliverti A, Cala SJ, Duranti R, Ferrigno G, Kenyon CM, Pedotti A, Scano G, Sliwinski P, Macklem PT, Yan S. Human respiratory muscle actions and control during exercise. J Appl Physiol (1985). 1997 Oct;83(4):1256-69. doi: 10.1152/jappl.1997.83.4.1256. PMID 9338435
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed